CLINICAL TRIAL: NCT01226745
Title: A Safety and Efficacy Extension Study of ONO-4641 (MSC2430913A) in Patients With Relapsing-Remitting Multiple Sclerosis
Brief Title: Phase 2 Extension Trial in Patients With Relapsing-Remitting Multiple Sclerosis (RRMS)
Acronym: DreaMS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Merck has decided to not pursue phase 3 development of ceralifimod (ONO-4641). The decision was not related to any safety and efficacy findings
Sponsor: EMD Serono (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry); Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ONO-4641POU007 (EMR200559-002); 2010-018705-11 (EudraCT Number)
Record Dates: First submitted 2010-10-19; First posted 2010-10-22 (Estimated); Results first posted 2016-07-12 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-06

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis; ONO-4641; MSC2430913A; Efficacy
MeSH Terms: conditions — Multiple Sclerosis | interventions — ceralifimod

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- ONO-4641 0.15 milligram (mg) - 0.15 mg (Experimental)
  Interventions: Drug: ONO-4641
- ONO-4641 0.10 mg - 0.10 mg (Experimental)
  Interventions: Drug: ONO-4641
- ONO-4641 0.05 mg - 0.05 mg (Experimental)
  Interventions: Drug: ONO-4641
- Placebo - ONO4641 0.15 mg (Experimental)
  Interventions: Drug: ONO-4641
- Placebo - ONO4641 0.10 mg (Experimental)
  Interventions: Drug: ONO-4641
- Placebo - ONO4641 0.05 mg (Experimental)
  Interventions: Drug: ONO-4641

INTERVENTIONS:
Drug: ONO-4641 — Subjects will be administered with ONO-4641 at a dose of 0.15 milligram (mg) in the core study will be administered with ONO-4641 0.15 mg in this extension study for a duration of 225 weeks.
  Other Names: MSC2430913A; Ceralifimod
  Arms: ONO-4641 0.15 milligram (mg) - 0.15 mg
Drug: ONO-4641 — Subjects will be administered with ONO-4641 at a dose of 0.10 mg in the core study will be administered with ONO-4641 0.10 mg in this extension study for a duration of 225 weeks.
  Other Names: MSC2430913A; Ceralifimod
  Arms: ONO-4641 0.10 mg - 0.10 mg
Drug: ONO-4641 — Subjects will be administered with ONO-4641 at a dose of 0.05 mg in the core study will be administered with ONO-4641 0.05 mg in this extension study for a duration of 225 weeks.
  Other Names: MSC2430913A; Ceralifimod
  Arms: ONO-4641 0.05 mg - 0.05 mg
Drug: ONO-4641 — Subjects will receive placebo in the core study will be administered with ONO-4641 0.15 mg in this extension study for a duration of 225 weeks.
  Other Names: MSC2430913A; Ceralifimod
  Arms: Placebo - ONO4641 0.15 mg
Drug: ONO-4641 — Subjects will receive placebo in the core study will be administered with ONO-4641 0.10 mg in this extension study for a duration of 225 weeks.
  Other Names: MSC2430913A; Ceralifimod
  Arms: Placebo - ONO4641 0.10 mg
Drug: ONO-4641 — Subjects will receive placebo in the core study will be administered with ONO-4641 0.05 mg in this extension study for a duration of 225 weeks.
  Other Names: MSC2430913A; Ceralifimod
  Arms: Placebo - ONO4641 0.05 mg

SUMMARY:
The objective of this active-drug Extension Study is to evaluate the continuing safety and efficacy of ONO-4641 (MSC2430913A) in subjects with relapsing-remitting multiple sclerosis (RRMS) who have completed an initial 26-week Core Study (ONO-4641POU006 [NCT01081782]).

ELIGIBILITY:
Inclusion Criteria:

* Completed 26 weeks of double-blind phase of Study ONO-4641POU006

Exclusion Criteria:

* Presence of any dermatological abnormalities during Study ONO-4641POU006 that could increase the risk of the patient developing a skin cancer

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 340 (Actual)
Dates: Start 2010-10; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — EMD Serono Inc., an affiliate of Merck KGaA, Darmstadt, Germany; Medical Responsible, Study Director — Ono Pharmaceutical Co. Ltd
Locations (70):
- United States (20):
  - Tucson Clinical Site 133, Tucson, Arizona
  - Aurora Clinical Site 132, Aurora, Colorado
  - Fort Collins Clinical Site 123, Fort Collins, Colorado
  - Fairfield Clinical Site 110, Fairfield, Connecticut
  - Ormond Beach Clinical Site 129, Ormond Beach, Florida
  - Sarasota Clinical Site 116, Sarasota, Florida
  - Northbrook Clinical Site 135, Northbrook, Illinois
  - Fort Wayne Clinical Site 111, Fort Wayne, Indiana
  - Indianapolis Clinical Site 121, Indianapolis, Indiana
  - Detroit Clinical Site 104, Detroit, Michigan
  - Farmington Hills Clinical Site 126, Farmington Hills, Michigan
  - Lebanon Clinical Site 115, Lebanon, New Hampshire
  - Albuquerque Clinical Site 106, Albuquerque, New Mexico
  - Rochester Clinical Site 108, Rochester, New York
  - Charlotte Clinical Site 125, Charlotte, North Carolina
  - Raleigh Clinical Site 103, Raleigh, North Carolina
  - Akron Clinical Site 112, Akron, Ohio
  - Philadelphia Clinical Site 120, Philadelphia, Pennsylvania
  - Knoxville Clinical Site 134, Knoxville, Tennessee
  - Round Rock Clinical Site 107, Round Rock, Texas
- Belgium (2):
  - Brugge Clinical Site 203, Bruges
  - La Louviere Clinical Site 201, La Louvière
- Canada (5):
  - Vancouver Clinical Site 131, Vancouver, British Columbia
  - Gatineau Clinical Site 114, Gatineau, Quebec
  - Greenfield park Clinical Site 109, Greenfield Park, Quebec
  - Montreal Clinical Site 101, Montreal, Quebec
  - Montreal Clinical Site 102, Montreal
- Czechia (3):
  - Olomouc Clinical Site 212, Olomouc
  - Pardubice Clinical Site 211, Pardubice
  - Praha 5 Clinical Site 213, Prague
- Germany (4):
  - Glessen Clinical Site 221, Glessen
  - Leipzig Clinical Site 229, Leipzig
  - Marburg Clinical Site 228, Marburg
  - Tubingen Clinical Site 226, Tübingen
- Athens Clinical Site 243, Athens, Greece
- Japan (9):
  - Kanto Region Clinical Site 404, Kanto
  - Kanto Region Clinical Site 405, Kanto
  - Kanto Region Clinical Site 406, Kanto
  - Kanto Region Clinical Site 409, Kanto
  - Kinki Region Clinical Site 401, Kinki
  - Kinki Region Clinical Site 407, Kinki
  - Kinki Region Clinical Site 408, Kinki
  - Tohoku Region Clinical Site 403, Tōhoku
  - Tohoku Region Clinical Site 410, Tōhoku
- Poland (8):
  - Bialystok Clinical Site 305, Bialystok
  - Czeladz Clinical Site 303, Czeladź
  - Gdansk Clinical Site 302, Gdansk
  - Katowice Clinical Site 309, Katowice
  - Krakow Clinical Site 307, Krakow
  - Lodz Clinical Site 306, Lodz
  - Plewiska Clinical Site 304, Plewiska
  - Warszawa Clinical Site 308, Warsaw
- Russia (8):
  - Kazan Clinical Site 333, Kazan'
  - Moscow Clinical Site 332, Moscow
  - Moscow Clinical Site 330, Moscow
  - Nizhniy Novgorod Clinical Site 321, Nizhny Novgorod
  - Novosibirsk Clinical Site 324, Novosibirsk
  - St. Petersburg Clinical Site 325, Saint Petersburg
  - Samara Clinical Site 329, Samara
  - Ufa Clinical Site 326, Ufa
- Spain (6):
  - Barcelona Clinical Site 252, Barcelona
  - Barcelona Clinical Site 253, Barcelona
  - Bilbao Clinical Site 255, Bilbao
  - Girona Clinical Site 254, Girona
  - Hospitalet de Llobregat Clinical Site 251, L'Hospitalet de Llobregat
  - Sevilla Clinical Site 256, Seville
- Ukraine (4):
  - Dnipropetrovsk Clinical Site 341, Dnipropetrovsk
  - Kyiv Clinical Site 344, Kyiv
  - Lviv Clinical Site 343, Lviv
  - Vinnytsya Clinical Site 342, Vinnytsia

REFERENCES:
- [Result] Effect of Ceralifimod (ONO-4641), a Sphingosine-1-Phosphate Receptor-1 and -5 Agonist, on Magnetic Resonance Imaging Outcomes in Patients with Multiple Sclerosis: Interim Results from the Extension of the DreaMS Study (P3.161) Amit Bar-Or, Frauke Zipp, Matthew Scaramozza, Timothy Vollmer, Bryan Due, Karthinathan Thangavelu, Tanya Fischer, and Krzysztof Selmaj April 8, 2014 82:10 Supplement P3.161; 1526-632X

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One Subject received 0.15 mg of ONO-4641 instead of placebo in error in the core trial and was subsequently re-randomized during the extension trial and received 0.10 mg of ONO-4641.This subject was not reported in the participant flow for the study.
Groups:
- ONO-4641 0.15 Milligram (mg) - 0.15 mg: Subjects who were administered with ONO-4641 at a dose of 0.15 mg in the core study were administered with ONO-4641 at a dose of 0.15 mg once daily in the extension study for a duration of 225 weeks.
- ONO-4641 0.10 mg - 0.10 mg: Subjects who were administered with ONO-4641 at a dose of 0.10 mg in the core study were administered with ONO-4641 at a dose of 0.10 mg once daily in the extension study for a duration of 225 weeks.
- ONO-4641 0.05 mg - 0.05 mg: Subjects who were administered with ONO-4641 at a dose of 0.05 mg in the core study were administered with ONO-4641 at a dose of 0.05 mg once daily in the extension study for a duration of 225 weeks.
- Placebo - ONO4641 0.15 mg: Subjects who were administered with placebo in the core study were administered with ONO-4641 at a dose of 0.15 mg once daily in the extension study for a duration of 225 weeks.
- Placebo - ONO4641 0.10 mg: Subjects who were administered with placebo in the core study were administered with ONO-4641 at a dose of 0.10 mg once daily in the extension study for a duration of 225 weeks.
- Placebo - ONO4641 0.05 mg: Subjects who were administered with placebo in the core study were administered with ONO-4641 at a dose of 0.05 mg once daily in the extension study for a duration of 225 weeks.
Period: Overall Study
Arm/Group | ONO-4641 0.15 Milligram (mg) - 0.15 mg | ONO-4641 0.10 mg - 0.10 mg | ONO-4641 0.05 mg - 0.05 mg | Placebo - ONO4641 0.15 mg | Placebo - ONO4641 0.10 mg | Placebo - ONO4641 0.05 mg
Started | 80 | 87 | 89 | 29 | 26 | 29
Completed | 63 | 71 | 69 | 24 | 22 | 24
Not Completed | 17 | 16 | 20 | 5 | 4 | 5
Not completed — Did not complete schedule of assessments | 8 | 3 | 6 | 0 | 0 | 1
Not completed — Lost to Follow-up | 2 | 6 | 6 | 1 | 1 | 2
Not completed — Death | 1 | 0 | 0 | 0 | 0 | 1
Not completed — Other | 6 | 7 | 8 | 4 | 3 | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis set consisted of all the enrolled subjects.
Groups:
- ONO-4641 0.15 mg - 0.15 mg: Subjects who were administered with ONO-4641 at a dose of 0.15 mg in the core study were administered with ONO-4641 at a dose of 0.15 mg once daily in the extension study for a duration of 225 weeks.
- Total: Total of all reporting groups
Arm/Group | ONO-4641 0.15 mg - 0.15 mg | ONO-4641 0.10 mg - 0.10 mg | ONO-4641 0.05 mg - 0.05 mg | Placebo - ONO4641 0.15 mg | Placebo - ONO4641 0.10 mg | Placebo - ONO4641 0.05 mg | Total
Number analyzed (Participants) | 80 | 87 | 89 | 29 | 26 | 29 | 340
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.3 (8.47) | 36.0 (8.64) | 38.2 (8.66) | 35.6 (9.59) | 37.0 (6.96) | 38.7 (9.48) | 36.9 (8.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 74 | 66 | 18 | 17 | 24 | 252
  Male | 27 | 13 | 23 | 11 | 9 | 5 | 88

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Clinically Significant Abnormal Vital Signs
Description: Vital signs included oral temperature, pulse, respiration rate and blood pressure (BP) (taken after 5 minutes in the sitting position). The abnormalities in vital signs were decided as clinically significant or not based on the clinical judgment of the investigator.
Time Frame: Baseline up to Week 255
Population: Safety analysis set consisted of all the enrolled subjects.
Measure: Number; unit: Subjects
Arm/Group | ONO-4641 0.15 mg - 0.15 mg | ONO-4641 0.10 mg - 0.10 mg | ONO-4641 0.05 mg - 0.05 mg | Placebo - ONO4641 0.15 mg | Placebo - ONO4641 0.10 mg | Placebo - ONO4641 0.05 mg
Number analyzed (Participants) | 80 | 87 | 89 | 29 | 26 | 29
Subjects | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Number of Gadolinium (Gd)-Enhanced Lesions
Description: Gd-enhanced lesions were obtained by magnetic resonance imaging (MRI) at each scheduled assessment visit over the study period. Extension study baseline is defined as the measurement most immediately prior to or on the day of the first dose day of extension study. End of treatment (EoT) lesion count is the average number of lesion counts per scan, calculated by dividing the sum of all lesion counts by number of scans during the extension treatment period. Early termination visit was recorded when the subject was early terminated from the study during the first 2.5 year period, while early termination 2 visit was recorded when the subject early terminated from the study during the additional 2 year period with delay. Extension study baseline is defined as the measurement most immediately prior to or on the day of the first dose day of extension study.Full Analysis Set (FAS) included all subjects who provided any post baseline efficacy data.
Time Frame: Baseline, Week 40, 52, 100, 148, early termination, Week 152, 200, early termination 2, Week 255 and end of treatment (5 years)
Population: FAS. "n" signifies the number of subjects analyzed for individual time point in the outcome measure.One randomized error subject was summarized in the sequence 0.15-0.15 as he received 0.15 in core study period and in the sequence Placebo-0.10 mg as he received 0.10 in the extension study period.
Measure: Mean (Standard Deviation); unit: Lesions
Arm/Group | ONO-4641 0.15 mg - 0.15 mg | ONO-4641 0.10 mg - 0.10 mg | ONO-4641 0.05 mg - 0.05 mg | Placebo - ONO4641 0.15 mg | Placebo - ONO4641 0.10 mg | Placebo - ONO4641 0.05 mg
Number analyzed (Participants) | 81 | 87 | 89 | 28 | 27 | 28
Lesions
  Baseline | 0.2 (0.57) | 0.0 (0.18) | 0.3 (0.65) | 2.7 (3.88) | 3.6 (10.46) | 1.6 (3.74)
  Week 40 (n=78, 84, 82, 28, 24, 25) | 0.2 (0.67) | 0.1 (0.62) | 0.4 (1.32) | 0.2 (0.42) | 0.3 (1.00) | 0.2 (0.50)
  Week 52 (n=77, 84, 77, 25, 24, 21) | 0.2 (0.86) | 0.2 (1.23) | 0.4 (0.93) | 0.2 (0.65) | 0.1 (0.34) | 0.4 (0.68)
  Week 100 (n=71, 73, 72, 22, 24, 18) | 0.1 (0.49) | 0.2 (0.76) | 0.4 (1.37) | 0.2 (0.53) | 0.1 (0.34) | 0.1 (0.47)
  Week 148 (n=61, 67, 68, 18, 22, 18) | 0.0 (0.22) | 0.1 (0.99) | 0.6 (1.85) | 0.0 (0.00) | 0.2 (0.66) | 0.1 (0.47)
  Early termination (n=16, 14, 13, 6, 3, 6) | 0.8 (2.76) | 0.1 (0.36) | 1.5 (4.68) | 0.2 (0.41) | 0.0 (0.00) | 0.5 (0.84)
  Week 152 (n=11, 10, 8, 4, 3, 6) | 0.2 (0.60) | 0.6 (0.97) | 2.5 (6.30) | 0.8 (1.50) | 0.0 (0.00) | 0.3 (0.82)
  Week 200 (n=20, 18, 21, 28, 27, 28) | 0.0 (0.00) | 0.5 (1.29) | 0.2 (0.89) | 0.0 (0.00) | 0.5 (1.22) | 0.0 (0.00)
  Early Termination 2 (n=58, 61, 60, 17, 21, 16) | 0.1 (0.34) | 0.2 (0.87) | 0.2 (0.38) | 0.1 (0.33) | 0.2 (0.51) | 0.4 (1.26)
  Week 255 (n=46, 48, 48, 16, 17, 13) | 1.1 (5.90) | 0.3 (1.01) | 0.4 (1.38) | 1.6 (3.90) | 0.2 (0.53) | 0.3 (0.85)
  End of treatment (n=80, 84, 85, 28, 24, 25) | 0.1 (0.39) | 0.2 (0.64) | 0.4 (0.93) | 0.2 (0.39) | 0.2 (0.53) | 0.3 (0.50)

3. Secondary Outcome: Change From Baseline in Lesion Volume at the End of the Treatment (EoT)
Description: Brain lesion volume was obtained by magnetic resonance imaging (MRI). Extension study baseline was defined as the measurement most immediately prior to or on the day of the first dose day of extension study. End of treatment (EOT) was defined as the last visit during the treatment period. Change from extension baseline to EOT = last treatment period value in extension study - extension baseline value.
Time Frame: Baseline, End of treatment (5 years)
Population: FAS included all subjects who provided any post baseline efficacy data.One randomized error subject was summarized in the sequence 0.15-0.15 as he received 0.15 in core study period and in the sequence Placebo-0.10 mg as he received 0.10 in the extension study period.
Measure: Mean (Standard Deviation); unit: Cubic centimeter (cc)
Arm/Group | ONO-4641 0.15 mg - 0.15 mg | ONO-4641 0.10 mg - 0.10 mg | ONO-4641 0.05 mg - 0.05 mg | Placebo - ONO4641 0.15 mg | Placebo - ONO4641 0.10 mg | Placebo - ONO4641 0.05 mg
Number analyzed (Participants) | 81 | 87 | 89 | 28 | 27 | 28
Cubic centimeter (cc) | -0.0264 (0.15483) | 0.0294 (0.11275) | 0.0197 (0.19925) | -0.4548 (0.96555) | -0.4465 (1.22881) | -0.1105 (0.36973)

4. Secondary Outcome: Percent Brain Volume Change (PBVC) From Baseline at the End of Treatment
Description: Brain volume was obtained by magnetic resonance imaging (MRI). Extension study baseline is defined as the measurement most immediately prior to or on the day of the first dose day of extension study. Brain volume changes very little over time. Hence, the PBVC at the end of treatment was calculated by adding up all the PBVC values from the scans performed during the extension treatment period.
Time Frame: Baseline and at end of treatment (Week 255)
Population: FAS included all subjects who provided any post baseline efficacy data. One randomized error subject was summarized in the sequence 0.15-0.15 as he received 0.15 in core study period and in the sequence Placebo-0.10 mg as he received 0.10 in the extension study period.
Measure: Mean (Standard Deviation); unit: Percent brain volume
Arm/Group | ONO-4641 0.15 mg - 0.15 mg | ONO-4641 0.10 mg - 0.10 mg | ONO-4641 0.05 mg - 0.05 mg | Placebo - ONO4641 0.15 mg | Placebo - ONO4641 0.10 mg | Placebo - ONO4641 0.05 mg
Number analyzed (Participants) | 81 | 87 | 89 | 28 | 27 | 28
Percent brain volume | -0.845 (0.8745) | -0.713 (0.8558) | -0.757 (0.7554) | -0.756 (0.8239) | -1.302 (0.9643) | -0.972 (0.8215)

5. Primary Outcome: Change From Baseline in Forced Expiratory Volume in One Second (FEV1) (Percent (%) Predicted Value)
Description: FEV1 was defined as the maximal volume of air exhaled in the 1st second of a forced expiration from a position of full inspiration. FEV1 was obtained from spirometry, performed before study treatment administration. Early termination visit was recorded when the subject was early terminated from the study during the first 2.5 year period, while early termination 2 visit was recorded when the subject early terminated from the study during the additional 2 year period with delay shall be defined.
Time Frame: Baseline, Week 40, 52, 76, 100, 124, 148, early termination, Week 152, 200, early termination 2, Week 255
Population: Safety analysis set consisted of all the enrolled subjects. Here "n" signifies the number of subjects analyzed for the individual time point in the outcome measure.
Measure: Mean (Standard Deviation); unit: Percentage of predicted value
Arm/Group | ONO-4641 0.15 Milligram (mg) - 0.15 mg | ONO-4641 0.10 mg - 0.10 mg | ONO-4641 0.05 mg - 0.05 mg | Placebo - ONO4641 0.15 mg | Placebo - ONO4641 0.10 mg | Placebo - ONO4641 0.05 mg
Number analyzed (Participants) | 80 | 87 | 89 | 29 | 26 | 29
Percentage of predicted value
  Week 40 (n=77, 83, 82, 29, 24, 24) | -0.227 (6.5379) | -0.741 (6.2026) | -0.062 (5.4947) | -1.500 (5.0115) | -1.555 (7.8424) | -1.146 (4.7952)
  Week 52 (n=74, 84, 77, 25, 24, 21) | -0.675 (7.7166) | -1.981 (6.8499) | -0.484 (6.0952) | -3.113 (5.4753) | -2.851 (6.7997) | -0.561 (5.5040)
  Week 76 (n=72, 78, 74, 24, 24, 21) | 1.148 (9.5950) | -2.352 (6.1152) | 0.650 (7.2084) | -1.574 (6.3645) | -2.300 (9.2869) | 2.657 (8.9280)
  Week 100 (n=68, 70, 72, 24, 24, 18) | -0.746 (8.3955) | -2.790 (8.2129) | -1.187 (7.8818) | -3.202 (6.7073) | -3.748 (8.5817) | -1.207 (7.7400)
  Week 124 (n=66, 70, 68, 21, 23, 18) | -0.795 (9.6531) | -2.003 (7.7998) | 0.197 (7.9068) | -2.178 (9.7656) | -1.968 (9.2415) | -0.874 (8.2237)
  Week 148 (n=59, 67, 68, 20, 21, 18) | -1.828 (10.8131) | -3.429 (8.4036) | -1.234 (6.5270) | -0.459 (9.0302) | -3.052 (9.4970) | -2.599 (10.3997)
  Early termination (n=16, 17, 13, 7, 3, 8) | -6.803 (6.7393) | 0.443 (6.0840) | -1.780 (11.6068) | -2.984 (13.8177) | -4.109 (21.4354) | 2.108 (8.1682)
  Week 152 (n=12, 12, 10, 4, 3, 8) | -3.786 (7.3297) | 4.515 (11.3809) | -1.725 (7.4166) | -11.929 (13.1156) | -11.525 (12.3316) | 2.688 (5.5468)
  Week 200 (n=18, 18, 19, 6, 6, 3) | -0.024 (8.0705) | -0.354 (12.8489) | -2.144 (8.3421) | -2.299 (8.2038) | -4.557 (13.3731) | 0.944 (7.8955)
  Early termination 2(n=56, 63, 63, 19, 20, 16) | -1.416 (9.4274) | -2.031 (10.6185) | -2.859 (9.6661) | -1.321 (8.7759) | -1.291 (10.4528) | -3.249 (11.5213)
  Week 255 (n=47, 48, 47, 17, 16, 13) | -0.368 (13.5515) | -1.374 (11.0920) | -0.027 (13.0574) | -0.209 (12.1999) | -2.377 (11.6511) | -0.963 (14.2975)

6. Primary Outcome: Change From Baseline in Forced Vital Capacity (FVC)
Description: FVC (% of predicted value) was the volume of air which was forcibly exhaled from the lungs after taking the deepest breath possible. Early termination visit was recorded when the subject was early terminated from the study during the first 2.5 year period, while early termination 2 visit was recorded when the subject early terminated from the study during the additional 2 year period with delay shall be defined.
Time Frame: Baseline, Week 40, 52, 76, 100, 124, 148, early termination, Week 152, 200, early termination 2, Week 255
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Percentage of predicted value
Arm/Group | ONO-4641 0.15 mg - 0.15 mg | ONO-4641 0.10 mg - 0.10 mg | ONO-4641 0.05 mg - 0.05 mg | Placebo - ONO4641 0.15 mg | Placebo - ONO4641 0.10 mg | Placebo - ONO4641 0.05 mg
Number analyzed (Participants) | 80 | 87 | 89 | 29 | 26 | 29
Percentage of predicted value
  Week 40 (n=77,83,82,29,24,24) | -0.123 (6.9868) | -1.000 (6.4060) | 0.921 (6.9931) | -1.593 (5.0520) | 1.554 (7.9727) | -0.423 (5.5244)
  Week 52 (n=74, 84, 77, 25, 24, 21) | -0.681 (6.1396) | -1.175 (6.1523) | 0.107 (7.7364) | -2.690 (5.2847) | -0.111 (6.2548) | -1.442 (6.8125)
  Week 76 (n=72, 78, 74, 24, 24, 21) | 1.397 (8.1634) | -1.906 (6.0432) | 1.828 (10.0612) | -2.487 (6.5830) | 0.568 (6.4530) | -0.707 (11.3657)
  Week 100 (n=68, 70, 72, 24, 24, 18) | -0.308 (7.9759) | -2.433 (6.6780) | 0.118 (7.8025) | -2.683 (4.9870) | -1.623 (8.3312) | -2.927 (7.8670)
  Week 124 (n=66, 70, 68, 21, 23, 18) | -0.794 (7.8392) | -2.246 (6.5967) | 0.890 (7.8545) | -2.582 (8.4640) | -0.487 (8.2776) | -1.821 (7.7421)
  Week 148 (n=59, 67, 68, 20, 21, 18) | -0.909 (6.7009) | -3.078 (6.6149) | 0.124 (7.7589) | -2.010 (7.8162) | -0.715 (6.7088) | -4.803 (9.3143)
  Early termination(n=16, 17, 13, 7, 3, 8) | -4.225 (8.2667) | -0.632 (5.1482) | 979.704 (3533.9625) | 0.278 (9.2002) | 0.459 (16.2506) | 2.813 (6.3216)
  Week 152 (n=12, 12, 10, 4, 3, 8) | -4.256 (7.4403) | -0.074 (6.8982) | -2.829 (7.0313) | -3.748 (9.0311) | -2.726 (17.6042) | -1.283 (9.7590)
  Week 200 (n=18, 18, 19, 6, 6, 3) | -0.316 (5.0212) | -3.057 (12.0551) | -1.590 (8.9426) | -1.109 (5.4668) | -1.152 (14.6922) | 4.287 (8.1537)
  Early termination (n=56, 63, 63, 19, 20, 16) | -0.033 (6.5169) | -1.952 (9.6157) | -0.903 (10.0341) | -1.593 (8.6842) | -0.892 (5.6941) | -4.731 (12.9422)
  Week 255 (n=47, 48, 47, 17, 16, 13) | -0.717 (8.1437) | -1.686 (10.4560) | 1.386 (13.9970) | -0.115 (13.4126) | -1.059 (10.2246) | -0.675 (11.1022)

7. Primary Outcome: Change From Baseline in Diffusing Capacity of Lung for Carbon Monoxide (DLCO)
Description: DLCO was one of the most clinically valuable tests of lung function. The DLCO measure the ability of the lungs to transfer gas from inhaled air to the red blood cells in pulmonary capillaries. Early termination visit was recorded when the subject was early terminated from the study during the first 2.5 year period, while early termination 2 visit was recorded when the subject was early terminated from the study during the additional 2 year period with delay. The values for the DLCO "% of predicted" was defined as the mean value of 2 test results that were within a 10% variability of each other.
Time Frame: Baseline, Week 40, 52, early termination, Week 152, 200, 255
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Percentage of predicted value
Arm/Group | ONO-4641 0.15 mg - 0.15 mg | ONO-4641 0.10 mg - 0.10 mg | ONO-4641 0.05 mg - 0.05 mg | Placebo - ONO4641 0.15 mg | Placebo - ONO4641 0.10 mg | Placebo - ONO4641 0.05 mg
Number analyzed (Participants) | 80 | 87 | 89 | 29 | 26 | 29
Percentage of predicted value
  Week 40 (n=22, 21, 16, 8, 9, 4) | 2.4 (13.16) | -1.0 (10.98) | -2.4 (17.36) | -5.3 (16.02) | -2.7 (10.61) | 3.3 (6.40)
  Week 52 (n=20, 19, 19, 8, 9, 5) | -3.7 (8.36) | -2.7 (10.74) | 0.8 (20.01) | -5.3 (11.56) | -4.8 (8.04) | 5.2 (6.34)
  Early termination (n=2, 1, 2, 3, 0, 0) | -6.5 (2.12) | -9.0 (NA) — Standard deviation is not evaluable as it is assessed only for 1 subject. | -43.0 (46.67) | -16.3 (12.58) | NA (NA) — Zero subjects were assessed for this measure. Hence, no data available. | NA (NA) — Zero subjects were assessed for this measure. Hence, no data available.
  Week 152 (n=3, 1, 2, 1, 0, 0) | -1.0 (1.00) | 11.0 (NA) — Standard deviation is not evaluable as it is assessed only for 1 subject. | 9.5 (3.54) | -14.0 (NA) — Standard deviation is not evaluable as it is assessed only for 1 subject. | NA (NA) — Zero subjects were assessed for this measure. Hence, no data available. | NA (NA) — Zero subjects were assessed for this measure. Hence, no data available.
  Week 200 (n=7, 5, 5, 2, 3, 2) | 3.0 (43.89) | 2.0 (12.85) | 35.8 (34.87) | 9.5 (28.99) | 25.0 (12.00) | 5.0 (9.90)
  Week 255 (n=14, 15, 12, 4, 6, 4) | 42.3 (40.41) | 21.0 (29.40) | 27.8 (37.38) | 5.8 (32.79) | 37.5 (40.78) | 16.3 (19.52)

8. Primary Outcome: Number of Subjects With Clinically Significant Abnormal Electrocardiogram (ECG) Measures
Description: The 12-lead ECG was recorded after the subject was in supine position for 5 minutes. ECGs were acquired on digital cardiographs. Abnormal findings were analyzed as clinically significant or not clinically significant as per the discretion of the study investigator.
Time Frame: Baseline up to Week 255
Population: Safety analysis set consisted of all the enrolled subjects.
Measure: Number; unit: Subjects
Arm/Group | ONO-4641 0.15 mg - 0.15 mg | ONO-4641 0.10 mg - 0.10 mg | ONO-4641 0.05 mg - 0.05 mg | Placebo - ONO4641 0.15 mg | Placebo - ONO4641 0.10 mg | Placebo - ONO4641 0.05 mg
Number analyzed (Participants) | 80 | 87 | 89 | 29 | 26 | 29
Subjects | 4 | 0 | 0 | 0 | 0 | 2

9. Primary Outcome: Number of Subjects With Clinically Significant Abnormal Ophthalmologic Examination
Description: Subjects underwent comprehensive ophthalmic examination (COE) including best corrected visual acuity (Snellen), manifest refractions, pupil examination, ocular motility, nystagmus, confrontation visual fields, Ishihara color plates, Amsler grid, and tonometry as well as a biomicroscopy slit lamp examination of the conjunctiva, cornea, anterior chamber, iris and lens; and a fundoscopic examination (with dilation) of the vitreous, optic nerve, retinal vessels, macula, and peripheral retina. Optical Coherence Tomography (OCT): Thicknesses of the macular retina and retinal nerve fiber layer at the optic nerve head in each eye was assessed by OCT using the fast macular thickness map scan and the fast retinal nerve fiber layer (RNFL) scan features, respectively. The abnormalities of the ophthalmologic examination was judged to be clinically significant or not as per the investigators discretion. The ophthalmologic examination was performed for both right eye (RE) and left eye (LE).
Time Frame: Baseline up to Week 255
Population: as for outcome 5
Measure: Number; unit: Subjects
Arm/Group | ONO-4641 0.15 mg - 0.15 mg | ONO-4641 0.10 mg - 0.10 mg | ONO-4641 0.05 mg - 0.05 mg | Placebo - ONO4641 0.15 mg | Placebo - ONO4641 0.10 mg | Placebo - ONO4641 0.05 mg
Number analyzed (Participants) | 80 | 87 | 89 | 29 | 26 | 29
Subjects
  COE: RE: Baseline (n=80, 87, 89, 29, 26,29) | 1 | 4 | 3 | 2 | 0 | 0
  COE: LE: Baseline (n=80, 87, 89, 29, 26, 29) | 0 | 4 | 3 | 2 | 0 | 0
  COE: RE: Week 40 (n=78, 81, 82, 25, 23, 24) | 2 | 2 | 2 | 1 | 0 | 0
  COE: LE: Week 40 (n=78, 81, 82, 25, 23, 24) | 5 | 1 | 2 | 1 | 0 | 0
  COE: RE: Week 52 (n=76, 83, 77, 26, 24, 21) | 0 | 2 | 4 | 1 | 0 | 0
  COE: LE: Week 52 (n=76, 83, 77, 26, 24, 21) | 2 | 2 | 3 | 1 | 0 | 0
  COE: RE: Week 76 (n=72, 79, 72, 24, 24, 21) | 1 | 2 | 4 | 1 | 0 | 1
  COE: LE: Week 76 (n=72, 79, 72, 24, 24, 21) | 3 | 2 | 5 | 1 | 0 | 1
  COE: RE: Week 100 (n=67, 72, 71, 24, 23, 18) | 2 | 2 | 0 | 1 | 0 | 0
  COE: LE: Week 100 (n=67, 72, 71, 24, 23, 18) | 5 | 1 | 1 | 1 | 0 | 0
  COE: RE: Week 124 (n=65, 69, 67, 20, 22, 18) | 2 | 2 | 3 | 1 | 0 | 0
  COE: LE: Week 124 (n=65, 69, 67, 20, 22, 18) | 2 | 2 | 1 | 1 | 1 | 0
  COE: RE: Week 148 (n=58, 66, 67, 19, 21, 18) | 2 | 2 | 3 | 1 | 0 | 0
  COE: LE: Week 148 (n=58, 66, 67, 19, 21, 18) | 3 | 3 | 4 | 1 | 0 | 0
  COE: RE: Early termination (n=15, 14, 16, 6, 2, 8) | 0 | 0 | 1 | 0 | 0 | 0
  COE: LE: Early termination (n=15, 14, 16, 6, 2, 8) | 1 | 0 | 1 | 0 | 0 | 0
  COE: RE: Week 152 (n=12, 11, 11, 3, 2, 9) | 0 | 0 | 2 | 0 | 0 | 0
  COE: LE: Week 152 (n=12, 11, 11, 3, 2, 9) | 1 | 0 | 1 | 0 | 0 | 0
  COE: RE: Week 174 (n=57, 61, 63, 17, 21, 15) | 0 | 2 | 4 | 1 | 0 | 0
  COE: LE: Week 174 (n=57, 61, 63, 17, 21, 15) | 2 | 2 | 2 | 1 | 0 | 0
  COE: RE: Week 200 (n=19, 18, 19, 5, 5, 4) | 0 | 1 | 0 | 1 | 0 | 0
  COE: LE: Week 200 (n=19, 18, 19, 5, 5, 4) | 0 | 1 | 0 | 1 | 0 | 0
  COE: RE: Week 225 (n=3, 2, 0, 0, 0, 0) | 0 | 0 | 0 | 0 | 0 | 0
  COE: LE: Week 225 (n=3, 2, 0, 0, 0, 0) | 0 | 0 | 0 | 0 | 0 | 0
  COE: RE: Early termination 2(n=50,56,62,19,21,16) | 1 | 2 | 2 | 1 | 0 | 0
  COE: LE: Early termination 2(n=50,56,62,19,21,16) | 1 | 2 | 3 | 1 | 0 | 0
  COE: RE: Week 255 (n=43, 42, 44, 16, 14, 13) | 1 | 0 | 3 | 1 | 0 | 0
  COE: LE: Week 255 (n=43, 42, 44, 16, 14, 13) | 1 | 0 | 3 | 1 | 0 | 0
  OCT: RE: Baseline (n=80, 87, 89, 29, 26, 29) | 4 | 2 | 4 | 1 | 0 | 1
  OCT: LE: Baseline (n=80, 87, 89, 29, 26, 29) | 4 | 1 | 2 | 1 | 0 | 1
  OCT: RE: Week 40 (n=76, 80, 81, 25, 23, 24) | 2 | 1 | 3 | 0 | 0 | 1
  OCT: LE: Week 40 (n=76, 80, 82, 25, 23, 24) | 2 | 1 | 3 | 1 | 0 | 1
  OCT: RE: Week 52 (n=74, 82, 74, 25, 22, 20) | 1 | 1 | 2 | 1 | 0 | 0
  OCT: LE: Week 52 (n=74, 82, 74, 25, 22, 20) | 1 | 1 | 2 | 2 | 0 | 0
  OCT: RE: Week 76 (n=69, 77, 72, 24, 24, 21) | 2 | 0 | 1 | 0 | 0 | 0
  OCT: LE: Week 76 (n=70, 77, 72, 24, 24, 21) | 2 | 0 | 1 | 2 | 0 | 0
  OCT: RE: Week 100 (n=66, 71, 70, 23, 23, 18) | 3 | 0 | 1 | 0 | 0 | 0
  OCT: LE: Week 100 (n=66, 71, 70, 23, 23, 18) | 2 | 0 | 1 | 2 | 0 | 0
  OCT: RE: Week 124 (n=64, 68, 66, 19, 21, 18) | 3 | 0 | 1 | 0 | 0 | 0
  OCT: LE: Week 124 (n=64, 68, 66, 19, 21, 18) | 2 | 1 | 1 | 1 | 0 | 0
  OCT: RE: Week 148 (n=57, 67, 67, 20, 21, 18) | 2 | 1 | 2 | 0 | 0 | 0
  OCT: LE: Week 148 (n=57, 67, 67, 20, 21, 18) | 2 | 1 | 2 | 1 | 0 | 0
  OCT: RE: Early termination (n=14, 15, 15, 8, 2, 8) | 0 | 0 | 1 | 1 | 0 | 1
  OCT: LE: Early termination (n=14, 15, 15, 8, 2, 8) | 0 | 0 | 1 | 1 | 0 | 1
  OCT: RE: Week 152 (n=12, 11, 10, 3, 2, 9) | 0 | 0 | 2 | 0 | 0 | 1
  OCT: LE: Week 152 (n=12, 11, 10, 3, 2, 9) | 0 | 0 | 0 | 0 | 0 | 1
  OCT: RE: Week 174 (n=57, 60, 63, 17, 21, 15) | 2 | 1 | 3 | 0 | 1 | 0
  OCT: LE: Week 174 (n=57, 60, 63, 17, 21, 15) | 3 | 1 | 2 | 1 | 1 | 0
  OCT: RE: Week 200 (n=18, 15, 20, 5, 5, 4) | 1 | 0 | 0 | 0 | 0 | 0
  OCT: LE: Week 200 (n=18, 15, 20, 5, 5, 4) | 0 | 0 | 0 | 1 | 0 | 0
  OCT: RE: Week 225 (n=2, 2, 0, 0, 0, 0) | 0 | 0 | 0 | 0 | 0 | 0
  OCT: LE: Week 225 (n=2, 2, 0, 0, 0, 0) | 0 | 0 | 0 | 0 | 0 | 0
  OCT:RE:Early termination 2(n=51, 55, 62,19,21,16) | 4 | 0 | 2 | 0 | 0 | 0
  OCT:LE:Early termination 2(n=51, 55, 62,19,21,16) | 2 | 0 | 1 | 1 | 0 | 0
  OCT: RE: Week 255 (n=43, 42, 41, 15, 14, 13) | 2 | 0 | 2 | 0 | 0 | 0
  OCT: LE: Week 255 (n=42, 42, 41, 15, 14, 13) | 2 | 0 | 1 | 1 | 0 | 0

10. Primary Outcome: Number of Subjects With Clinically Significant Abnormalities in Dermatological Examination
Description: A whole body examination, paying particular attention to identify precancerous or cancerous lesions was done by a dermatologist and based on the clinical judgment of the dermatologist the abnormalities were categorized as clinically significant or clinically not significant. Early termination visit was recorded when the subject was early terminated from the study during the first 2.5 year period, while early termination 2 visit was recorded when the subject early terminated from the study during the additional 2 year period with delay shall be defined.
Time Frame: Baseline up to end of the treatment, assessed up to Week 255
Population: Safety analysis set consisted of all the enrolled subjects.
Measure: Number; unit: Subjects
Arm/Group | ONO-4641 0.15 mg - 0.15 mg | ONO-4641 0.10 mg - 0.10 mg | ONO-4641 0.05 mg - 0.05 mg | Placebo - ONO4641 0.15 mg | Placebo - ONO4641 0.10 mg | Placebo - ONO4641 0.05 mg
Number analyzed (Participants) | 80 | 87 | 89 | 29 | 26 | 29
Subjects
  Baseline | 1 | 0 | 3 | 1 | 0 | 1
  Week 40 | 1 | 2 | 3 | 1 | 0 | 0
  Week 52 | 3 | 4 | 3 | 0 | 0 | 1
  Week 76 | 4 | 4 | 3 | 2 | 1 | 0
  Week 100 | 5 | 2 | 2 | 2 | 1 | 1
  Week 124 | 6 | 7 | 2 | 2 | 1 | 1
  Week 148 | 3 | 5 | 1 | 2 | 0 | 2
  Early termination | 0 | 1 | 0 | 1 | 0 | 0
  Week 152 | 0 | 1 | 0 | 0 | 0 | 0
  Week 174 | 2 | 1 | 1 | 0 | 1 | 1
  Week 200 | 1 | 1 | 0 | 1 | 0 | 0
  Early termination 2 | 1 | 0 | 0 | 1 | 0 | 1
  Week 255 | 1 | 0 | 0 | 0 | 0 | 0

11. Primary Outcome: Number of Subjects With Treatment Emergent Adverse Events (TEAEs), Serious TEAEs, TEAEs Leading to Death and TEAEs Leading to Discontinuation
Description: An Adverse Event (AE) was defined as any new untoward medical occurrences/worsening of pre-existing medical condition without regard to possibility of causal relationship. A Serious Adverse Event (SAE) was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect. TEAEs were defined as the AEs that occur between first dose of study drug administration and 35 days after the last dose of study drug administration that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: From the first dose of study drug administration up to 35 days after the last dose of study drug administration, assessed up to 5 years
Population: Safety analysis set consisted of all the enrolled subjects.
Measure: Number; unit: Subjects
Arm/Group | ONO-4641 0.15 mg - 0.15 mg | ONO-4641 0.10 mg - 0.10 mg | ONO-4641 0.05 mg - 0.05 mg | Placebo - ONO4641 0.15 mg | Placebo - ONO4641 0.10 mg | Placebo - ONO4641 0.05 mg
Number analyzed (Participants) | 80 | 87 | 89 | 29 | 26 | 29
Subjects
  TEAEs | 75 | 85 | 82 | 27 | 22 | 29
  Serious TEAEs | 16 | 12 | 21 | 5 | 9 | 11
  TEAEs leading to death | 1 | 0 | 0 | 0 | 0 | 1
  TEAEs leading to discontinuation | 6 | 6 | 7 | 3 | 2 | 6

ADVERSE EVENTS:
Time Frame: From the administration of study medication up to the final study visit, assessed up to 5 years
Arm/Group | ONO-4641 0.15 Milligram (mg) - 0.15 mg | ONO-4641 0.10 mg - 0.10 mg | ONO-4641 0.05 mg - 0.05 mg | Placebo - ONO4641 0.15 mg | Placebo - ONO4641 0.10 mg | Placebo - ONO4641 0.05 mg
Serious Adverse Events (participants affected / at risk) | 16/80 | 12/87 | 21/89 | 5/29 | 9/26 | 11/29
Other Adverse Events (participants affected / at risk) | 67/80 | 80/87 | 72/89 | 21/29 | 21/26 | 27/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ONO-4641 0.15 Milligram (mg) - 0.15 mg (N=80) | ONO-4641 0.10 mg - 0.10 mg (N=87) | ONO-4641 0.05 mg - 0.05 mg (N=89) | Placebo - ONO4641 0.15 mg (N=29) | Placebo - ONO4641 0.10 mg (N=26) | Placebo - ONO4641 0.05 mg (N=29)
Multiple sclerosis relapse (Nervous system disorders) | 4 | 8 | 11 | 1 | 6 | 6
Cerebral infarction (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Paraparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Appendicitis perforated (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Encephalitic infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Lymphangitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Meningitis aseptic (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1
Blood human chorionic gonadotropin increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Colonic polyp (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Peritonitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Connective tissue disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Autism spectrum disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Mania (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Chemical poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Pelvic prolapse (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Uterine polyp (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Female sterilisation (Surgical and medical procedures) | 2 | 0 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
External ear inflammation (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0
Retinal detachment (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Retinal tear (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Venous insufficiency (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ONO-4641 0.15 Milligram (mg) - 0.15 mg (N=80) | ONO-4641 0.10 mg - 0.10 mg (N=87) | ONO-4641 0.05 mg - 0.05 mg (N=89) | Placebo - ONO4641 0.15 mg (N=29) | Placebo - ONO4641 0.10 mg (N=26) | Placebo - ONO4641 0.05 mg (N=29)
Nasopharyngitis (Infections and infestations) | 18 | 21 | 22 | 3 | 8 | 7
Upper respiratory tract infection (Infections and infestations) | 14 | 21 | 15 | 4 | 5 | 6
Urinary tract infection (Infections and infestations) | 7 | 16 | 13 | 2 | 4 | 6
Bronchitis (Infections and infestations) | 12 | 8 | 8 | 2 | 0 | 0
Oral herpes (Infections and infestations) | 2 | 9 | 7 | 0 | 5 | 0
Pharyngitis (Infections and infestations) | 3 | 9 | 6 | 2 | 0 | 3
Sinusitis (Infections and infestations) | 8 | 6 | 7 | 0 | 2 | 0
Influenza (Infections and infestations) | 3 | 6 | 5 | 1 | 1 | 3
Gastroenteritis viral (Infections and infestations) | 4 | 2 | 6 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 3 | 3 | 1 | 1 | 0 | 2
Cystitis (Infections and infestations) | 3 | 1 | 2 | 0 | 2 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 2 | 1 | 0 | 2
Onychomycosis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 2
Headache (Nervous system disorders) | 13 | 13 | 13 | 7 | 5 | 2
Multiple sclerosis relapse (Nervous system disorders) | 4 | 9 | 12 | 1 | 7 | 7
Dizziness (Nervous system disorders) | 4 | 8 | 3 | 2 | 1 | 1
Hypoaesthesia (Nervous system disorders) | 5 | 3 | 5 | 2 | 0 | 2
Migraine (Nervous system disorders) | 5 | 4 | 3 | 0 | 2 | 0
Muscle spasticity (Nervous system disorders) | 1 | 5 | 2 | 0 | 1 | 1
Paraesthesia (Nervous system disorders) | 4 | 2 | 1 | 0 | 0 | 1
Sciatica (Nervous system disorders) | 0 | 2 | 3 | 1 | 0 | 2
Tremor (Nervous system disorders) | 1 | 2 | 1 | 0 | 0 | 2
Memory impairment (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 11 | 8 | 12 | 1 | 5 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 8 | 6 | 1 | 3 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 | 4 | 8 | 3 | 0 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 4 | 5 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 3 | 5 | 0 | 0 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 3 | 1 | 1 | 3
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 | 2 | 6 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2 | 1 | 0
Alanine aminotransferase increased (Investigations) | 8 | 8 | 12 | 6 | 3 | 6
Gamma-glutamyltransferase increased (Investigations) | 7 | 9 | 9 | 4 | 3 | 5
Aspartate aminotransferase increased (Investigations) | 3 | 4 | 4 | 3 | 0 | 4
Activated partial thromboplastin time (Investigations) | 2 | 3 | 2 | 0 | 2 | 1
Blood cholesterol increased (Investigations) | 2 | 2 | 3 | 0 | 2 | 1
Blood creatine phosphokinase increased (Investigations) | 3 | 1 | 4 | 0 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 8 | 10 | 4 | 1 | 2 | 1
Nausea (Gastrointestinal disorders) | 8 | 7 | 4 | 0 | 0 | 3
Abdominal pain upper (Gastrointestinal disorders) | 3 | 5 | 4 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 4 | 2 | 4 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 4 | 4 | 1 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 4 | 2 | 2 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 5 | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 2
Contusion (Injury, poisoning and procedural complications) | 3 | 8 | 3 | 1 | 2 | 5
Fall (Injury, poisoning and procedural complications) | 4 | 3 | 3 | 1 | 2 | 3
Procedural pain (Injury, poisoning and procedural complications) | 4 | 4 | 1 | 1 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 4 | 4 | 1 | 0 | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 0 | 4 | 1 | 0 | 2 | 2
Joint sprain (Injury, poisoning and procedural complications) | 2 | 2 | 1 | 0 | 1 | 2
Foreign body in eye (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2 | 0
Insomnia (Psychiatric disorders) | 4 | 10 | 6 | 2 | 1 | 2
Depression (Psychiatric disorders) | 4 | 7 | 5 | 1 | 0 | 4
Anxiety (Psychiatric disorders) | 7 | 2 | 2 | 1 | 0 | 2
Acne (Skin and subcutaneous tissue disorders) | 5 | 5 | 5 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 7 | 4 | 1 | 0 | 0 | 2
Increased tendency to bruise (Skin and subcutaneous tissue disorders) | 2 | 7 | 0 | 1 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 3 | 2 | 1 | 0 | 1 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 5 | 1 | 0 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 0 | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 6 | 8 | 2 | 2 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 | 3 | 2 | 1 | 1 | 2
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 5 | 0 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 2 | 0 | 0 | 0
Fatigue (General disorders) | 6 | 10 | 9 | 1 | 3 | 3
Pyrexia (General disorders) | 3 | 4 | 6 | 0 | 2 | 0
Conjunctivitis (Eye disorders) | 2 | 1 | 6 | 0 | 1 | 0
Retinal disorder (Eye disorders) | 1 | 2 | 2 | 2 | 0 | 0
Blepharospasm (Eye disorders) | 2 | 0 | 0 | 0 | 0 | 2
Conjunctival hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 2 | 0
Hypertension (Vascular disorders) | 6 | 2 | 3 | 1 | 4 | 5
Vertigo (Ear and labyrinth disorders) | 5 | 5 | 5 | 0 | 1 | 1
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3 | 5 | 1 | 2 | 2
Seasonal allergy (Immune system disorders) | 3 | 5 | 6 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 5 | 2 | 1 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 1 | 5 | 0 | 1 | 1
Lymphopenia (Blood and lymphatic system disorders) | 1 | 3 | 0 | 0 | 2 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0 | 1 | 2 | 0 | 0

LIMITATIONS AND CAVEATS:
Company has decided to not pursue phase 3 development of ceralifimod (ONO-4641). The decision was not related to any safety and efficacy findings.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other